CLINICAL TRIAL: NCT01635023
Title: A Phase I, Single-center, Randomized, Open-label, Crossover Study to Compare the White (Current Phase II) and Blue (Planned Phase III) Capsule Formulations of AZD6244 Hyd-Sulfate in Healthy Male Subjects
Brief Title: A Randomized, Open Label Study to Compare the Current Phase II and Planned Phase III Capsule Formulation of AZD6244
Acronym: AZD6244Formula
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D1532C00066
Record Dates: First submitted 2012-06-25; First posted 2012-07-06 (Estimated); Last update posted 2012-10-25 (Estimated); Status verified 2012-10

CONDITIONS: Healthy Volunteers
Keywords: Phase I; healthy volunteers; AZD6244; pharmacokinetics; AUC; Cmax; tmax; AUC(0-t)
MeSH Terms: interventions — AZD 6244

ARMS (3):
- AZD6244 white capsule (Experimental): 75mg AZD6244 white (current Phase II) capsule
  Interventions: Drug: AZD6244 Dosing Period 1; Drug: AZD6244 Dosing Period 2; Drug: AZD6244 Dosing Period 3
- AZD6244 blue capsule (Experimental): 75mg AZD6244 blue (planned Phase III) capsule
  Interventions: Drug: AZD6244 Dosing Period 1; Drug: AZD6244 Dosing Period 2; Drug: AZD6244 Dosing Period 3; Drug: AZD6244 Dosing Period 4
- AZD6244 solution (Experimental): 35mg AZD6244 oral solution
  Interventions: Drug: AZD6244 Dosing Period 1; Drug: AZD6244 Dosing Period 2; Drug: AZD6244 Dosing Period 3

INTERVENTIONS:
Drug: AZD6244 Dosing Period 1 — Treatment A, B, or C depending on randomization assignment
  Other Names: AZD6244
Drug: AZD6244 Dosing Period 2 — Treatment A, B, or C depending on randomization assignment
  Other Names: AZD6244
Drug: AZD6244 Dosing Period 3 — Treatment A, B, or C depending on randomization assignment
  Other Names: AZD6244
Drug: AZD6244 Dosing Period 4 — Treatment B
  Other Names: AZD6244
  Arms: AZD6244 blue capsule

SUMMARY:
Study in Healthy Males to Compare the White and Blue Formulations of AZD6244.

DETAILED DESCRIPTION:
A Phase I, Single-center, Randomized, Open-label, Crossover Study to Compare the White (Current Phase II) and Blue (Planned Phase III) Capsule Formulations of AZD6244 Hyd-Sulfate in Healthy Male Subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers aged 18 to 55 BMI between 18 and 30 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg, inclusive Calculated creatinine clearance (CRCL) greater than 50 mL/min usin gthe Cockcroft-Gault formula

Exclusion Criteria:

* History or presence of gastrointestinal, hepatic, or renal disease or any other condition know to interfere with absorption, distribution, metabolism, or exertion of drugs.
* Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody, or HIV.
* Any clinically important abnormalities in rhythm, conduction, or morphology of the resting dECG and any clinically important abnormalities in the 12-lead dECG that suggest a cardiac, metabolic or other noncardiac condition.
* Current or past history of central serous retinopathy or retinal vein thrombosis, intraocular pressure greater than 21 mmHg or uncontrolled glaucoma Known or suspected history of drug abuse, current smokes or those who have smoked or used nicotine-containing products within the previous 3 months

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2012-07; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
AUC for AZD6244 administered as a single dose of white (current Phase II) capsule formulation | Measured at appropriate time-points until end of treatment peiod, approximately 24 days
Cmax for AZD6244 administered as a ingle dose of white (current Phase II) capsule formulation | Measured at appropriate time-points until end of treatment peiod, approximately 24 days
AUC for AZD6244 administered as a single dose of blue (planned Phase III) capsule formulation | Measured at appropriate time-points until end of treatment peiod, approximately 24 days
Cmax for AZD6244 administered as a single dose of blue (planned Phase III) capsule formulation | Measured at appropriate time-points until end of treatment peiod, approximately 24 days

SECONDARY OUTCOMES:
Frequency and severity of adverse events | Measured throughout the study and for a7 days after the last dose, approximately 29 days
AUC for AZD6244 administered as a single dose of oral solution formulation | Measured at appropriate time-points until end of treatment peiod, approximately 24 days
Cmax for AZD6244 administered as a single dose of oral solution formulation | Measured at appropriate time-points until end of treatment peiod, approximately 24 days

CONTACTS AND LOCATIONS:
Overall Officials: Ian Smith, MEDICAL SCIENCE DIRECTOR, Study Director — AstraZeneca; Eleanor Lisbon, MD, Principal Investigator — Quintiles, Inc.
Locations (1):
- Reseatch Site, Overland Park, Kansas, United States

REFERENCES:
- [Derived] Tomkinson H, McBride E, Martin P, Lisbon E, Dymond AW, Cantarini M, So K, Holt D. Comparison of the Pharmacokinetics of the Phase II and Phase III Capsule Formulations of Selumetinib and the Effects of Food on Exposure: Results From Two Randomized Crossover Trials in Healthy Male Subjects. Clin Ther. 2017 Nov;39(11):2260-2275.e1. doi: 10.1016/j.clinthera.2017.08.022. Epub 2017 Oct 4. PMID 28985960